CLINICAL TRIAL: NCT05320562
Title: Effect of Kinesio Taping and Sham Taping on Knee Function in Patients With Knee Osteoarthritis: Randomized Clinical Trial
Brief Title: Effect of Kinesio Taping and Sham Taping in Knee Osteoarthritis
Acronym: OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuanianSportsU-8
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis
Keywords: kinesiotaping; functional mobility; physiotherapy; knee pain
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Participants underwent 3 exercise sessions for 60 minutes each. Exercise program was created to improve range of motion and muscle strength. Participants executed active exercise in lying, sitting, and standing positions, isometric exercise, exercise with resistance band. All exercises were repeated 12 times in 3 sets and depending on the capacity of the subject. Breaks between sets 10 sec.
- Sham taping (Sham Comparator): Participants underwent 3 exercise sessions for 60 minutes each. Exercise program was created to improve range of motion and muscle strength. Participants executed active exercise in lying, sitting, and standing positions, isometric exercise, exercise with resistance band. All exercises were repeated 12 times in 3 sets and depending on the capacity of the subject. Breaks between sets 10 sec.
  Interventions: Procedure: Sham taping
- Kinesio taping (Experimental): Participants underwent 3 exercise sessions for 60 minutes each. Exercise program was created to improve range of motion and muscle strength. Participants executed active exercise in lying, sitting, and standing positions, isometric exercise, exercise with resistance band. All exercises were repeated 12 times in 3 sets, 10 s breaks between sets.
  Interventions: Procedure: Kinesio taping

INTERVENTIONS:
Procedure: Kinesio taping — Additionally, they received kinesio taping application for 7 days. Blue color kinesio tape (manufactured by "Theraband®", USA) was used. Kinesio taping was done by experienced physiotherapist with 5 years of experience. Two Y shape bands were applied for lymphatic taping and to improve anterior upper leg muscle function (lymphatic correction and muscle correction techniques were integrated together).
  Then two I shape bands (75-100% tension) were applied above the patella tendon and medial/lateral collateral ligaments in order to improve mechanoreceptor stimulation, proprioception and knee stability.
  Arms: Kinesio taping
Procedure: Sham taping — Additionally, they received sham (placebo) taping: usual white patch was applied to the painful knee for 7 days. The technique of taping used was the same as in kinesiotaping group, but without stretching.
  Arms: Sham taping

SUMMARY:
The prevalence of knee osteoarthritis has been increasing in recent decades as the number of obese people has increased. Various interventions are used to improve the functional condition of patients, but it is still not clear which one is most effective. The primary aim of this study was to determine and compare the effects of kinesio taping and sham taping on the knee functional mobility.

DETAILED DESCRIPTION:
The investigators assigned 30 adult participants (26 women, 4 men; mean age 58,1±3,9 yrs) from Lithuania. Participants were assigned to one of three groups: control group (CON) (n = 10), sham taping + exercise (STE) (n = 10), and kinesio taping + exercise (KTE) group (n = 10). Participants performed all necessary tests according to the study protocol one week before the intervention. A second set of tests was performed one week after the intervention. The intervention duration was 1 week. Exercise, sham and kinesio taping were applied by Physical Therapist. All the study groups did exercise training.

ELIGIBILITY:
Inclusion Criteria:

* clinical and radiography diagnosis of osteoarthritis of the knee joint
* patients with different degrees of severity of the knee osteoarthritis
* consent to participate in the study.

Exclusion Criteria:

* rheumatoid arthritis
* systemic connective tissue disease
* knee joint oedema
* surgery intervention in recent 6 months
* wearing of knee braces
* skin problems
* previous total or partial knee replacement surgery
* inability to perform physical examination tests
* oncology
* use of medications, infection
* previous experience of kinesio taping intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Knee Pain at 1 week | Baseline and after 7 days
  was evaluated using the Visual Analogue Pain Scale (VAS). Participants were asked to report "current" pain intensity. A higher score indicates greater pain intensity: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
Change from Baseline Range of Motions at 1 week | Baseline and after 7 days
  A goniometer was used to measure the flexion and extension of the knee joint. The initial position of the subject is prone lying, the axis of goniometer is placed on the lateral femoral epicondyle. The stationary part of goniometer is placed along the lateral midline of the thigh, the reference point being the greater trochanter of femur. The moving part of goniometer is placed along the midline of the lower leg, the reference point being the lateral ankle.
Change from Baseline Muscle Strength at 1 week | Baseline and after 7 days
  Manual muscle strength testing. The strength of knee flexion and extension was evaluated (Cuthbert, & Goodheart, 2007). The classic 5-point manual muscle strength assessment system is used to determine muscle strength. If for some reason participant could not perform the full range of motion, then the muscle strength test is performed at the possible amplitude.
Change from Baseline Walking Speed at 1 week | Baseline and after 7 days
  A 10-meter straight line was marked in the start and finish points. The subject had to stand 2 meters in front of the start line, after the signal participant was told to walk at his/her own speed until he/she was 2 meters behind the finish line. The timer was turned on when the patient crossed the start line and stopped when he/she crossed the finish line. The test was performed 5 times and the average calculated. Time was recorded in seconds and converted to meters per second (Master et al., 2021).
Change from Baseline Functional Mobility at 1 week | Baseline and after 7 days
  Initial position was participant sitting on the chair. The patient had to get up from the chair, walk three meters to the marked line, turn around 180 degrees, and return to the chair, and sit down on the chair. During the test, the person must wear normal footwear and use all means of movement normally required. The test was performed 5 times and the average of 5 tests was calculated. The height of the chair used was 46 cm and the test time was recorded in seconds (Alghadir et al., 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania